CLINICAL TRIAL: NCT00604071
Title: Sensitivity of the Home Macular Perimeter (HMP) in the Detection of Visual Field Abnormalities in Patients With Choroidal Neovascularization (CNV) Secondary to Age Related Macular Degeneration (AMD)- PILOT Study
Brief Title: Sensitivity of the Home Macular Perimeter (HMP)
Acronym: HMP
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Other Study IDs: HMP-V4; 20071801
Record Dates: First submitted 2008-01-10; First posted 2008-01-29 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Age Related Macular Degeneration; Choroidal Neovascularization
Keywords: HMP, CNV, PHP, HPHP, AMD
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: subjects with AMD related lesions: New onset (up to 60 days) non-treated CNV

SUMMARY:
estimate the sensitivity of the HMP test in identifying visual field functional defects in subjects with CNV secondary to AMD

DETAILED DESCRIPTION:
The HMP device is intended to aid patients in identifying their visual abnormalities and in addition to their own symptoms or Amsler grid use and aid in their prompt referral to eye care professional examination so clinical diagnosis can be made. As such the goal of the clinical plan is to demonstrate that patients who have CNV do demonstrate visual field abnormalities when tested with the HMP

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to sign a consent form and participate in the study
* subjects with AMD related lesions: New onset (up to 60 days) non-treated CNV
* Age >50 years
* VA with habitual correction >20/200 in study eye
* Familiar with computer usage

Exclusion Criteria:

* Evidence of macular disease other than AMD or glaucoma in the study eye
* Presence of any significant media opacity that precludes a clear view of the macular area as identified in the study eye by biomicroscopy, CFP, or FA
* Any non-macular related ocular surgery performed within 3 months prior to study entry in the targeted eye
* Inability to tolerate intravenous FA
* Participation in another study with the exclusion of AREDS study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 62 completed subjects with new choroidal neovascularization AMD in at least one eye
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
estimate the sensitivity of the HMP test in identifying visual field functional defects in subjects with CNV secondary to AMD based on PRC grading of color stereo photographs and Stereoscopic fluorescein angiogram | 3 month

SECONDARY OUTCOMES:
Estimate the sensitivity of the HMP in identifying visual field functional defects in subjects with CNV secondary to AMD based in cases where both graders, prior to any adjudication process determined the presence of CNV | 3 month
Estimate the sensitivity of the HMP in identifying visual field functional defects in subjects with CNV secondary to AMD based on cases where both graders, prior to any adjudication process, and biomicroscopic finding determined the presence of CNV | 3 Month
Estimate the sensitivity of the HMP in identifying visual field functional defects in subjects with CNV secondary to AMD determined on biomicroscopy | 3 month
Estimate the sensitivity of the Amsler grid test in identifying functional changes in subjects with CNV secondary to AMD based on PRC grading of color stereo photographs and fluorescein angiograms. | 3 month
Estimate the sensitivity of the HMP test in identifying visual field functional defects in subjects with CNV secondary to AMD for each of three classifications of CNV lesions (occult, minimally classic and predominantly classic). | 3 month
Estimate the sensitivity of the HMP test in identifying visual field functional defects in subjects with CNV secondary to AMD which were either minimally classic or occult and where the physician elected to treatment over observation | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bressler, Prof., Principal Investigator — JHMC
Locations (10):
- United States (10):
  - Central Florida Retina Institute, Lakeland, Florida
  - Retina care specialists, Palm Beach Gardens, Florida
  - International Eye Center, Tampa, Florida
  - Center for Retina & Macular Disease, Winter Haven, Florida
  - Edina Retina Consultants, Edina, Minnesota
  - Retina Vitreous Center, New Brunswick, New Jersey
  - Foxman Foxman & Margolis, Northfield, New Jersey
  - Harkness Eye institute, West New York, New Jersey
  - Charlotte Eye Ear Nose & Throat, Charlotte, North Carolina
  - Virginia Retina Center, Leesburg, Virginia

REFERENCES:
- See also: sponsor web site — http://www.notalvision.com